CLINICAL TRIAL: NCT06631144
Title: Improving Health Equities for Hispanic/Latino Families Living With Dementia by Validating a Spanish-language Caregiver-Enabled Care Program (CECP) in PACE Participants
Brief Title: A Spanish-language Caregiver-Enabled Care Program
Acronym: CECP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ceresti Health, Inc. (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CER-2024-111-001; 1R43AG088143-01 (NIH)
Record Dates: First submitted 2024-08-27; First posted 2024-10-08 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Dementia; Dementia Alzheimers; Alzheimer Disease; Caregiver; Caregiver Burden
Keywords: Digital Health Intervention; Spanish
MeSH Terms: conditions — Dementia; Alzheimer Disease; Caregiver Burden

STUDY DESIGN:
Intervention Model Description: A single-arm feasibility study to test a non-medical digital health intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Caregiver-Enabled Care Group (Experimental): Caregiver participants will receive Ceresti's Caregiver-Enabled Care Program. (CECP) is a 6-month non-medical digital program that promotes the wellness of family caregivers, and increases their knowledge, skills and confidence ("activation") in caring for a loved one with dementia. CECP delivers personalized health education, access to resources, proactive coaching, personalized support, and remote monitoring via a dedicated tablet that is shipped to the caregiver's home.
  Interventions: Behavioral: Spanish-language Caregiver-Enabled Care Program (CECP)

INTERVENTIONS:
Behavioral: Spanish-language Caregiver-Enabled Care Program (CECP) — CECP is a nonmedical digital population health intervention to support and engage family caregivers of persons with dementia. CECP consists of digital content, including health education videos and tutorials, that is delivered to caregivers on a dedicated tablet based on their specific needs. Caregivers are supported by a proactive human coach who provides support, access to resources, and performs risk mitigation measures as necessary. Alerts are shared with providers and/or care management teams via a data hub that makes it easy to track, manage and resolve alerts. CECP is delivered over a 6-month period via a dedicated tablet that is shipped to the caregiver's home at no cost to the caregiver or person with dementia. This study's CECP is in Spanish.

SUMMARY:
The purpose of the study is to develop and test the feasibility of a nonmedical digital health intervention, the Spanish-language Caregiver-Enabled Care Program (CECP), with Spanish-speaking caregivers of persons with dementia (PWD). CECP is a nonmedical digital population health intervention that provides personalized education, proactive 1:1 human coaching, and remote monitoring, all delivered via a dedicated tablet shipped to the caregiver's home at no cost to the caregiver or PWD. For this study, the investigators are recruiting 135 patient/caregiver dyads.

DETAILED DESCRIPTION:
For Hispanic/Latino families in the United States (U.S.), care for a loved one with dementia is provided largely by family caregivers. Evidence-based resources that support and engage family caregivers are critical to improving care and outcomes for persons living with dementia and improving the wellness of their family caregiver. However, access to these vital resources is limited for Hispanic/Latino families in the U.S. To address health disparities in dementia care for Hispanic/Latino families in the U.S., the investigators are developing an approach for deploying the proven Caregiver-Enabled Care Program (CECP) to Spanish-speaking caregivers of patients with dementia. For this study, the investigators will enroll 135 Spanish-speaking family caregiver/dementia-patient dyads living in the U.S. who are participants in a Program for All-Inclusive Care for the Elderly (PACE) or dementia support network or provider. Participation for each caregiver enrolled in the study involves engaging in the Spanish-language CECP for 6 months. The overall duration of the research project is 12 months.

At the conclusion of the study, the investigators expect to show that the highly- scalable approach using Artificial Intelligence (AI) plus human validation provides a Spanish-language CECP that can achieve comparable engagement of the proven English-language CECP. The investigators will measure differences in how Spanish-speaking caregivers engage in education, coaching, and assessments compared to the engagement of English-speaking caregivers. Understanding these differences will allow the investigators to explore potential cultural differences in user engagement and inform future optimization of the program. This Phase 1 Small Business Innovation Research (SBIR) study is supported by the National Institute On Aging (NIA) of the National Institutes of Health (NIH) under Award Number R43AG088143.

ELIGIBILITY:
Patient/Caregiver Dyad Inclusion Criteria

Patient Inclusion Criteria:

* Is a participant of a Program of All-Inclusive Care for the Elderly (PACE) or dementia support network or provider in the United States
* Identifies as Hispanic/Latino
* Has a Spanish-speaking familial caregiver (spouse, adult child, other family member, or friend) that is willing and able to participate in all aspects of this study
* Has a diagnosis of dementia
* Consents to participate in study, or has an Authorized Representative that consents

Caregiver Inclusion Criteria:

• Is a Spanish-speaking family caregiver (spouse, adult child, other family member, friend) providing care/support for the person with dementia

* Is an adult aged 18 or older
* Primary language is Spanish. Able to speak, read, and write Spanish
* Consents to participate in the study

Exclusion Criteria:

• Patient plans to disenroll from the PACE program or dementia support network or provider in in less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2024-12-04 (Actual); Primary Completion 2026-01-22 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
Longitudinal Engagement | From the date of enrollment in the program until the last assessment, assessed up to 6 months.
  Longitudinal Engagement for this study is assessed as the month-to-month continuation rate of Spanish-speaking caregivers enrolled in the CECP.
Intensity of Engagement | From the date of enrollment in the program until the last assessment, assessed up to 6 months.
  Intensity of Engagement for this study is assessed as the average weekly engagement time of enrolled Spanish-speaking caregivers in education, coaching and assessment of the CECP.

SECONDARY OUTCOMES:
Centers for Disease Control and Prevention (CDC) Healthy Days Measure (Spanish version) | From the date of enrollment until the last monthly assessment, assessed every month up to 6 months
  Centers for Disease Control and Prevention (CDC) Healthy Days Measure evaluates participants' health status over the past 30 days. For most questions, 0 days indicates the best health status, and 30 days indicates the worst health status. Higher scores on the Centers for Disease Control and Prevention (CDC) Healthy Days Measure generally indicate worse outcome, reflecting more days of poor physical and mental health. Additionally, participants identify their major health problem, indicate whether it limits daily living, and specify the level of assistance needed for personal care and routine activities by selecting one response from a provided list.
Caregiver Activation Scale (in Spanish) | From the date of enrollment until the last monthly assessment, assessed every month up to 6 months
  Custom question developed by Ceresti to measure increase in caregiver knowledge, skills and confidence. Higher scores on the Caregiver Activation Scale indicate better outcome.
Loneliness Scale (in Spanish) | From From the date of enrollment until the last monthly assessment, assessed every month up to 6 months
  Custom questions developed by Ceresti to measure feelings of loneliness experienced in the past 30 days. Higher scores on the Loneliness Scale indicate worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Soenksen, Principal Investigator — CEO
Locations (1):
- Ceresti Health, Carlsbad, California, United States

IPD SHARING:
Plan to Share IPD: No
De-identified, aggregated, summarized data will be made available for sharing.

DOCUMENTS (1):
  • Informed Consent Form (2024-09-27): https://cdn.clinicaltrials.gov/large-docs/44/NCT06631144/ICF_000.pdf